CLINICAL TRIAL: NCT03091348
Title: Subcutaneous Testosterone Therapy in Men Compared to Intramuscular Testosterone Therapy in Men
Brief Title: Subcutaneous vs. Intramuscular Testosterone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Men's Health Boston (Other)
Responsible Party: Principal Investigator, Dr. Abraham Morgentaler, Director, Men's Health Boston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MHB023
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Testosterone Deficiency; Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone; testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SQ - IM (Experimental): Subcutaneous testosterone injection followed by intramuscular testosterone injection
  Interventions: Drug: Testosterone
- IM - SQ (Experimental): Intramuscular testosterone injection followed by subcutaneous testosterone injection
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone cypionate injection
  Other Names: Testosterone cypionate; Testosterone injection

SUMMARY:
In this randomized, cross-over study 20 subjects who are undergoing testosterone (T) therapy for the treatment of T deficiency will receive both subcutaneous testosterone therapy and intramuscular testosterone therapy. One group will receive a SQ injection followed by an IM injection and one group will receive an IM injection followed by a SQ injection. The primary objective of this study is to measure testosterone concentration in men after these two treatment routes and determine if there are any significant differences due to modes of administration. Endpoints will include total serum testosterone and calculated free testosterone. A questionnaire will also be administered to assess overall patient experience with each route of administration.

DETAILED DESCRIPTION:
Subjects planning to initiate testosterone treatment via injection at MHB will be consented into the study. Upon enrollment in the study, the randomization will be completed for each subject.

Blood collection will occur before each injection. Subjects will rate pain on the Likert scale following each injection. After treatment with the first mode of T administration (SQ or IM depending on randomization), subjects will come in for blood draws 3 days and 7 days following the injection. Two weeks after the initial injection, subjects will come in for treatment with the second mode of T administration (SQ or IM depending on randomization). Subjects will come in for blood draws 3 days and 7 days following the second injection. Two weeks after the second injection, subjects will complete an end of study assessment with an Investigator and will complete a survey assessing their satisfaction with treatment. Subjects will likely continue testosterone therapy at Men's Health Boston after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, write, and understand English
* Age greater than or equal to 18
* Diagnosed with testosterone deficiency
* Pre-enrollment testosterone concentration of less than 350 ng/dL
* Planning to initiate testosterone treatment at MHB
* Willing to be followed at MHB for at least one month
* Willing to provide informed consent for this study

Exclusion Criteria:

* Previous exposure to exogenous T, clomiphene citrate, or other Selective Estrogen Receptor Modulators, unless off therapy for at least 12 weeks
* American Urological Association Prostate Symptom score of 15 or greater or significant prostatic symptoms
* History of carcinoma, tumors or induration of the prostate or the male mammary gland, including suspicion thereof
* Pre-enrollment serum PSA more than 4 ng/ml
* Serious psychiatric disease or uncontrolled medical illness, as suspected from the history or clinical examination
* Used any sex hormones or steroidal anabolic drug supplements within 28 days before pre-enrollment testosterone collection or at any time throughout the study
* Incapable of giving informed consent or complying with the protocol

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston, Harvard Medical School
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SQ - IM | IM - SQ
Started | 2 | 2
Completed | 0 | 1
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants analyzed is 0 and 1 due to loss to follow up
Groups:
- SQ-IM: Subcutaneous testosterone injection followed by intramuscular testosterone injection
  Testosterone: Testosterone cypionate injection
- IM-SQ: Intramuscular testosterone injection followed by subcutaneous testosterone injection
  Testosterone: Testosterone cypionate injection
- Total: Total of all reporting groups
Arm/Group | SQ-IM | IM-SQ | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: loss to follow up
  years |  | 44 (0) | 44 (0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: loss to follow up caused only 1 subject to be analyzed
  Participants
    Female | 0 | 0 | 0
    Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: loss to follow up
  Participants
    American Indian or Alaska Native |  | 0 | 0
    Asian |  | 0 | 0
    Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Black or African American |  | 0 | 0
    White |  | 1 | 1
    More than one race |  | 0 | 0
    Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
Estradiol (E2) [Number; unit: pg/ml] — Population: loss to follow up
  pg/ml |  | 24.5 | 24.5
Human Follicle Stimulating Hormone (hFSH) [Number; unit: miu/ml] — Population: loss to follow up
  miu/ml |  | 3.5 | 3.5
Hemophagocytic lymphohistiocytosis(hLH) [Number; unit: miu/ml] — Population: loss to follow up
  miu/ml |  | 3 | 3
Sex hormone binding globulin(SHBG) [Number; unit: nmol/l] — Population: loss to follow up
  nmol/l |  | 27.3 | 27.3
Testosterone [Number; unit: ng/dl] — Population: loss to follow up
  ng/dl |  | 317.1 | 317.1

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of Serum Total Testosterone Concentration
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7"
Population: loss to follow up
Measure: Number; unit: ng/dl
Groups:
- "SQ": Subcutaneous testosterone injection Testosterone: Testosterone cypionate injection
- "IM": Intramuscular testosterone injection Testosterone: Testosterone cypionate injection
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
ng/dl
  visit 2 | NA — design of the study is cross over, with only 1 subjects | 1043.6
  visit 3 | NA — design of the study is cross over, with only 1 subjects | 785.7
  visit 4 | 203.5 | NA — design of the study is cross over, with only 1 subjects
  vist 5 | 1367.9 | NA — design of the study is cross over, with only 1 subjects
  visit 6 | 980.8 | NA — design of the study is cross over, with only 1 subjects
  visit 7 | 144.7 | NA — design of the study is cross over, with only 1 subjects

2. Primary Outcome: Change in Levels of Serum Calculated Free T Concentration
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Last visit ( Visit 7)"
Population: loss to follow up
Measure: Number; unit: ng/dL
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
ng/dL | 0.84 | 14.74

3. Secondary Outcome: Change in Levels of Serum Estradiol
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7"
Population: loss to follow up
Measure: Number; unit: pg/mL
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
pg/mL
  visit 2 | NA — cross over study design | 70.03
  visit 3 | NA — cross over study design | 52.00
  visit 4 | 30.06 | NA — cross over study design
  visit 5 | 45.12 | NA — cross over study design
  visit 6 | 64.74 | NA — cross over study design
  visit 7 | 25.99 | NA — cross over study design

4. Secondary Outcome: Change in Levels of Serum LH
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7"
Population: loss to follow up
Measure: Number; unit: miu/ml
Groups:
- "IM": Intramuscular testosterone injection Testosterone : Testosterone cypionate injection
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
miu/ml
  visit 2 | NA — cross over study design | 0.4
  visit 3 | NA — cross over study design | 0.3
  visit 4 | 0.2 | NA — cross over study design
  visit 5 | 0.04 | NA — cross over study design
  visit 6 | 0.1 | NA — cross over study design
  visit 7 | 0.4 | NA — cross over study design

5. Secondary Outcome: Change in Levels of Serum FSH
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7"
Population: loss to follow up
Measure: Number; unit: miu/ml
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
miu/ml
  visit 2 | NA — cross over study design | 1.3
  visit 3 | NA — cross over study design | 0.4
  visit 4 | 0.2 | NA — cross over study design
  visit 5 | 0.1 | NA — cross over study design
  visit 6 | 0.05 | NA — cross over study design
  visit 7 | 0.3 | NA — cross over study design

6. Secondary Outcome: Change in Levels of Serum SHBG
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7"
Population: loss to follow up
Measure: Number; unit: nmol/l
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
nmol/l
  visit 2 | NA — cross over study design | 25.5
  visit 3 | NA — cross over study design | 22
  visit 4 | 27.8 | NA — cross over study design
  visit 5 | 24.8 | NA — cross over study design
  visit 6 | 22.9 | NA — cross over study design
  visit 7 | 20.7 | NA — cross over study design

7. Secondary Outcome: Change in Level of Serum PSA
Description: Blood samples measured by Beckman assays and equipment.
Time Frame: "Last visit (Visit 7)"
Population: loss to follow up
Measure: Number; unit: ng/mL
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
ng/mL | 0.25 | 0.02

8. Secondary Outcome: Change in Levels of Whole Blood Hematocrit
Description: Blood samples measured by Quest assays and equipment.
Time Frame: "Last visit (Visit 7)"
Population: loss to follow up
Measure: Number; unit: g/dL
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 1 | 1
g/dL | NA — insufficient number of participants with event/measures. | 1.9

9. Secondary Outcome: Change in Low Testosterone Questionnaire Responses
Description: Answers recorded at baseline, 2 weeks, up to 4 weeks. Scale is 1-5 (strongly disagree to strongly agree) Lower scores are better
Time Frame: after last vist #7
Population: loss to follow up
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in International Prostate Symptom Scores
Description: Answers recorded at baseline, 2 weeks, up to 4 weeks.
  Scale 0-35, from Mild to Severe Lower score is better
Time Frame: after last vist #7
Population: loss to follow up
Arm/Group | "SQ" | "IM"
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE were monitored/assessed at each study visit.
Description: An adverse event is defined as any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom, or disease temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research. Include the type and duration of the follow-up of subjects after adverse events.
Groups:
- SQ Testosterone: Subcutaneous testosterone injection Testosterone: Testosterone cypionate injection
- IM Testosterone: Intramuscular testosterone injection Testosterone: Testosterone cypionate injection
Arm/Group | SQ Testosterone | IM Testosterone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03091348/Prot_SAP_000.pdf